CLINICAL TRIAL: NCT01067430
Title: Comparison of the Effect of Etoricoxib and Diclofenac on Early Morning Activity in Rheumatoid Arthritis.
Brief Title: Comparison of the Effect of Etoricoxib and Diclofenac on Early Morning Activity in Rheumatoid Arthritis (RA)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr David Walker, Principal Investigator, Northumbria Healthcare NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IISP 35166
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Etoricoxib; Diclofenac; Pain; Stiffness
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Etoricoxib; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib 90 mg (Active Comparator): Subject will take Etoricoxib 90 mg for 14 days
  Interventions: Drug: Etoricoxib
- Diclofenac (Active Comparator): Film coated tablet 50 mgs given three times a day for 14 days
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Etoricoxib — Film coated tablet, 90 mg taken once a day for 14 days
  Other Names: Arcoxia
  Arms: Etoricoxib 90 mg
Drug: Diclofenac — Enteric coated tablet 50 mg given three times a day for 14 days
  Other Names: Voltarol
  Arms: Diclofenac

SUMMARY:
The purpose of this study is to explore the effect of Etoricoxib compared to Diclofenac on physical activity in RA subjects with early morning pain and stiffness.

DETAILED DESCRIPTION:
Rheumatoid Arhthitis (RA) is a chronic inflammatory condition characterised by prolonged morning stiffness. Anti-inflammatory medication is effective in relieving the pain and stiffness associated with this inflammation. By having a long half-life, Etoricoxib has a simple once daily dosing regime and the long action overnight should mean that patients experience more effective relief of symptoms first thing in the morning compared to shorter half life medication such as Diclofenac. The activity of people can be measured using the NuMact monitor which has been validated against observation and for use in RA . As the data is logged in real time it is possible to extract the periods of activity at the start of the day when morning stiffness will be maximal. It counts the number and vigour of steps.

This can be used to give a measure of total ambulatory activity but in this instance we are interested primarily in the vigour of step first thing in the morning. The vigour of the steps (trunk deceleration on heel strike) is a measure of how easily and quickly a subject is walking. We would expect this to be markedly reduced in people with RA during their period of "morning stiffness".

This is a study is of a randomised crossover design. The aim is to recruit 20 subjects suffering from Rheumatoid Arthritis. 20 has been chosen as a suitable number to show the effects of the two drugs and allow design of a definitive study. All participants will be tolerant of conventional NSAIDs.

All subjects will be given patient information sheets at least 24 hours before the first visit. They will be allowed time to read the information sheet and given the opportunity to ask further questions if they wish during the pre-baseline week.

The first visit is the baseline visit during which informed consent will be taken by the Chief Investigator, all of the inclusion and exclusion criteria will be checked to ensure the subject still meets the criteria. A history of NSAID use will also be taken to ensure subject tolerance of the drug. Quality of life Questionnaires will be administered during this visit, they will consist of the:

Health Assessment Questionnaire (HAQ) which assesses dressing, arising, eating, walking, hygiene, reach, grip and common activities. For each of these categories, patients report the amount of difficulty they have in performing two or three specific activities. There are 4 possible responses; without ANY difficulty; with SOME difficulty; with MUCH difficulty; UNABLE to do.

Pain VAS and Fatigue VAS The visual analog scale (VAS fatigue) is a horizontal line; 100 mm in length, self-administered by the patient in order to rate pain from 0 "no fatigue" to 100 "worst possible fatigue".

DAS28 is a measure of disease activity in rheumatoid arthritis (RA). The score is calculated by a mathematical formula, which includes the number of tender and swollen joints (out of a total of 28), the erythrocyte sedimentation rate (ESR, a blood marker of inflammation). A DAS28 score greater than 5.1 implies active disease, less than 3.2 well controlled disease, and less than 2.6 remission.

A physical examination by the Chief Investigator will also take place at this visit and concomitant medication and any adverse events occurring since receiving the patient information leaflet will be recorded.

Assessments will be done at baseline and after 2 weeks of treatment with each anti-inflammatory. At the baseline visit subjects will have a 48 hr run-in period where they will be allocated placebo. During this time a 24 hr recording using the NuMact Ambulatory device wll be taken. This has been included so that treatment effect vs placebo can be recorded which would strengthen the final analysis and findings. The NuMact ambulatory activity monitor will be used to assess spontaneous ambulatory activity.

After the 48 hr period the first arm of the study will commence and subjects will be randomly allocated to receive either Etoricoxib 90 mg once a day or Diclofenac 50 mg three times a day, which will be prescribed for 2 weeks. At the end of this period (visit 3), a further NuMact reading will take place and disease status will be assessed using the DAS 28, HAQ VAS Pain and VAS Fatigue. A home visit will take place to remove the NuMact device with the patient's consent. This has been written into the protocol because a second reading could take place should the reading fail at visit 3. At visit 5 the patient will return to the hospital to start the second arm of treatment where they will cross over to either Etoricoxib 90 mg tonce a day or Diclofenac 50 mg three times a day. They will be prescribed this medication for two weeks and at visit 6 another NuMact recording will take place and disease status will be assessed using the DAS 28, HAQ VAS Pain and VAS Fatigue. With the patient's consent, the device will be removed after 24 hrs at the patient's home.

Physical examination will be carried out at the baseline visit and at visits 3 and 6. It could be carried out at any time during the study period if considered appropriate by the physician.

Concomitant medication and therapy and adverse events will be recorded by the Investigator at each study visit.

A follow-up phone call will be undertaken 2 weeks after the final visit as a safety measure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years and over.
* Subjects who are NSAID tolerant.
* Subjects with a clinical diagnosis of rheumatoid arthritis.
* Subjects who are willing to complete QOL questionnaires.
* Written informed consent

Exclusion Criteria:

* Co-occurrence of other disabling conditions in addition to rheumatoid arthritis likely to warrant the persistent use of escape analgesia.
* Subjects who have received an intra-articular or muscular steroid injection within 3 months of study entry or in whom such treatment is planned within the study period.
* Subjects scheduled for elective surgery of the disease site or any other elective major surgery which would fall within the study period.
* Severe respiratory impairment.
* Clinically significant hepatic or renal dysfunction, subjects whose LFTs and serum creatinine is outside normal recognized limits.
* Subjects with convulsive disorders, head injury, shock, reduced level of consciousness of uncertain origin, intracranial lesions or increased intracranial pressure.
* Subjects with a known allergy or hypersensitivity to NSAIDs.
* Subjects with unstable gastro-intestinal complications or disease.
* Subjects who currently abuse alcohol or drugs, or have a recent history of alcohol or drug abuse, or who in the Investigator's opinion, have previously demonstrated drug-seeking behaviour.
* Subjects who are currently participating in another clinical research study involving a new chemical entity or who have participated in a clinical study within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
To explore the effect of Etoricoxib compared to Diclofenac on physical activity in RA subjects with Early morning pain and stiffness. | After 14 days of treatment
  Subjects will be asked to complete a visual analogue scale to record pain and stiffness and activity will be recorded with the Numact devise

CONTACTS AND LOCATIONS:
Overall Officials: David J Walker, MD, Principal Investigator — Northumbria Healthcare NHS Foundation Trust
Locations (1):
- Northumbria Healthcare NHS Foundation Trust, North Shields, Tyne and Wear, United Kingdom